CLINICAL TRIAL: NCT02164877
Title: A Randomized, Controlled Study of Soluble Dietary Fiber on Bacterial Translocation in Adults Patients With Crohn's Disease
Brief Title: Effect of Soluble Dietary Fiber on Bacterial Translocation in Crohn's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Not enough participants enrolled
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Jianfeng Gong, Associate professor, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pectin-2014
Record Dates: First submitted 2014-06-13; First posted 2014-06-17 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Crohn's Disease
Keywords: Dietary fiber
MeSH Terms: conditions — Crohn Disease | interventions — Pectins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pectin (Experimental): Patients allocated to experiment group will receive standard enteral nutrition formula(Fresubin) supplemented with 15g pectin each day for 4 weeks.
  Interventions: Drug: pectin
- control (Placebo Comparator): Patients allocated to control group will receive standard enteral nutrition formula(Fresubin) for 4 weeks
  Interventions: Drug: pectin

INTERVENTIONS:
Drug: pectin — Patients allocated to experiment group will receive 15g pectin each day
  Other Names: soluble dietary fiber

SUMMARY:
The purpose of this study is to evaluate the effect of soluble dietary fiber on bacterial translocation and mucosal immunology in patients with Crohn's disease.

DETAILED DESCRIPTION:
Bacterial translocation (BT) is a proposed mechanism of CD. Microorganisms can be cultured from 18-48% of draining mesenteric lymph nodes from CD patients. A breakdown in barrier function in "late stage" CD has been observed in patients requiring surgery. In addition, it was found that BT influences the response to biological therapy and clinical relapse in CD. Therefore, reducing BT may be of therapeutic importance in treatment for CD.

The role of soluble dietary fiber in Crohn's disease (CD) is still inconclusive. Population based studies have shown that long-term intake of dietary fiber is associated with lower risk of CD. However, meta-analysis did not show benefit in inducing or maintaining remission. In addition, the possible mechanism of dietary fiber on CD is still unclear.

The rationale relates to the beneficial effects of fiber may be due to the production of the fiber metabolites short-chain fatty acids (SCFAs), particularly butyrate. Dietary substrates may modify the commensal microbiota or their metabolites or enhance epithelial barrier function. Recently, it was found that dietary fiber metabolites SCFA is regulatory of mucosal regulatory T cells. The current study is to examine the impact of dietary fiber on bacterial translocation,intestinal luminal microbiology, and mucosal immunology in CD patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >=17 years with diagnosis of CD for at least 3 months defined by histology or radiology
* ileocolonic non-penetrating disease
* Moderate active CD with CDAI 250-450
* CRP level over normal range
* Stable CD therapy with a total steroid dose not exceeding 10mg prednisolone or equivalent for 4 weeks

Exclusion Criteria:

* Infection with enteric pathogen
* Usage of probiotics, antibiotics, or prebiotics within the last month
* Change in dose of oral steroids or 5-ASA within the last 4 weeks or AZA or MTX in the last 3 months
* Dose of steroids exceeds 10 mg prednisolone per day or equivalent
* Infusion of IFX or any alternative biological therapy within the last 3 months
* Use of rectal 5-ASA or steroids within the last 2 weeks.
* Imminent need for surgery or presence of severe disease (CDAI >450)
* Pregnancy or lactation
* Short bowel syndrome or subtotal/total colectomy
* Pure anal disease and previous proctocolectomy
* Significant hepatic, renal, endocrine, respiratory, neurological or cardiovascular disease as determined by the principal investigator
* History of cancer with a disease-free state of less than two years
* Patients with penetrating disease or small bowel lesion only.

Ages: 17 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2014-06; Primary Completion 2017-05 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
bacteria translocation in MLN, mesenteric fat and peripheral blood | 4 weeks after treatment
  Bacterial translocation to mesenteric lymph nodes (MLN),mesenteric fat and peripheral blood during laparotomy before surgical mobilization, as determined by DGGE.

SECONDARY OUTCOMES:
change of fecal bacteriology | baseline, week 4
  fecal microbiology before and 4 weeks after pectin treatment, as determined by DGGE
change of fecal SCFA | baseline, week 4
  fecal short chain fatty acid (SCFA) levels before and 4 weeks after treatment, as determined by HPLC.
clinical response | up to 4 weeks after treatment
  the percentage of patients achieving a clinical response (fall in CDAI of >=70 points) at week 4.
change of mucosal Treg numbers | baseline, week 4
  mucosal Treg（FoxP3+CD4+）cell number before and after treatment,as determined by immunofluorescence
adverse events | up to 4 weeks after treatment
  gastrointestinal symptoms(borborygmi,flatulence,abdominal pain,diarrhea etc)

CONTACTS AND LOCATIONS:
Overall Officials: Jianfeng Gong, MD, Principal Investigator — Department of general surgery,Jinling hospital
Locations (1):
- Department of Generay Surgery, Jinling hosptal, Medical School of Nanjing University, Nanjing, Jiangsu, China